CLINICAL TRIAL: NCT00656591
Title: An Evaluation of the Cost-Effectiveness of Community-Based Participatory Interventions for Pregnant Women in Nepal to Reduce Fetal and Infant Mortality, and to Improve Fetal Growth and Cognitive Development in Infancy.
Brief Title: Community-Based Interventions for Infant Health in Nepal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Responsible Party: R&D Office, Institute of Child Health
Other Study IDs: 04PC01
Record Dates: First submitted 2006-12-22; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Child Mortality
Keywords: Child mortality, Nepal, Community, care practices
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

INTERVENTIONS:
Drug: Methotrexate — Methotrexate

SUMMARY:
An Evaluation of the Cost-Effectiveness of Community-Based Participatory Interventions for Pregnant Women in Nepal to Reduce Fetal & Infant Mortality and to Improve Fetal Growth & Cognitive Development in Infancy

ELIGIBILITY:
Inclusion Criteria:

* mothers, community health volunteers

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 48 village development committee areas
Sampling Method: Probability Sample
Enrollment: 192000 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
neonatal mortality rates | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Costello, Dr, Principal Investigator — Institute of Child Health
Locations (1):
- International Child Health, ICH, London, United Kingdom